CLINICAL TRIAL: NCT00734006
Title: Cortico-cortical Connectivity During Midazolam Sedation in Humans; a TMS/EEG Study
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0018
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: Cortico-cortical; connectivity; Transcranial; Magnetic; Stimulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the proposed research is to measure the effect of drug-induced sedation on the functional connectivity between brain regions as indicated by EEG signal transmission within the human brain. The results of this study will help to identify the neurophysiological correlates of changes in conscious experience that occur during drug-induced sedation.

DETAILED DESCRIPTION:
In the proposed experiments cortical areas will be stimulated using low frequency, low-amplitude transcranial magnetic stimulation (TMS) in healthy human subjects during wakefulness and during drug-induced responsive sedation and unresponsive sedation. Simultaneously, high-density electroencephalography (Hd-EEG) will be recorded to evaluate the temporal and spatial characteristics of evoked responses and induced rhythms over the cortex.

ELIGIBILITY:
Inclusion Criteria:

* Healthy right-handed men
* Aged 18-35
* Non-smokers
* No metallic implants

Exclusion Criteria:

* Younger than 18 or over the age of 35.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy right-handed men aged 18-35 who do not smoke or have any metallic implants may be eligible for this study.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Defining the neurophysiological conditions that are necessary for conscious experience. | Immediate

SECONDARY OUTCOMES:
Understanding the neurophysiological correlates of conditions associated with restricted conscious experience such as sedation and anesthesia. | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pearce, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States